CLINICAL TRIAL: NCT03372031
Title: Active Versus Passive Piano Intervention for Dexterity in Older Adults: A Randomized Controlled Trial
Brief Title: The Effectiveness of Piano Therapy vs. Piano Listening on Manual Dexterity in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Westminster College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SeylerCapstone2017
Record Dates: First submitted 2017-12-08; First posted 2017-12-13 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Aging; Manual Dexterity; Piano Therapy
Keywords: Music Supported Therapy; plasticity; multisensory integration; bimanual coupling; auditory feedback; dexterity; piano therapy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized members of dyads (formed by residential treatment facility personnel) in to therapy order conditions. Two weeks piano therapy for one while the other listened followed by two week in reversed roles. Half the participants played first and listened second and the other half did the reverse.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active-Passive (Experimental): Active Piano training (8 sessions in two weeks) followed by listening to piano training (8 sessions in 2 weeks) (Passive condition)
  Interventions: Behavioral: Piano training (Active); Behavioral: Piano Training (Passive)
- Passive-Active (Experimental): Passive piano training listening (8 sessions in two weeks) followed by active piano training (8 sessions in two weeks)
  Interventions: Behavioral: Piano training (Active); Behavioral: Piano Training (Passive)

INTERVENTIONS:
Behavioral: Piano training (Active) — Piano Curriculum. Participants were all trained on one of four 88-key pianos located in the assisted living facility. Piano instructors were 6 undergraduate Music Education and Music Performance majors. Each lesson of the week had a different focus: right and left hands separately, bimanually coupled, and bimanually uncoupled (Loehrer et al., 2016). Each week of the module had a different focus as well: notes played one step apart, notes played multiple steps apart (intervals), and tones played together (two-note chords) (van Vugt et al., 2016; Villeneuve et al., 2014). Each session began with skill exercises and ended with learning a simple, recognizable song. Two participants with extensive piano experience progressed to playing duets with the instructor and hymns out of a hymnal after mastery of the study curriculum. These training protocols were based on those of Schneider and colleagues' 2007 study.
  Other Names: Piano Training (Passive)
Behavioral: Piano Training (Passive) — Participants listened to their research partner complete 8 active piano training sessions across 2 weeks.

SUMMARY:
Does active piano practice help recover hand dexterity in older adults, or does social interaction and music-listening alone affect motor performance? Researchers hypothesized improved dexterity after active piano playing, but not after passive piano listening. 15 residents of a retirement community were partnered together and completed 2 two-week piano training modules. In module 1, one partner played piano exercises and songs while the other listened. In module 2, partners switched roles. The Purdue Pegboard Test and Box and Block Test assessed fine and gross motor dexterity, before, between, and after the training modules. A repeated measures ANOVA showed a main effect of time on overall fine and gross motor function, but there was no main effect of playing versus listening. Results did not support the hypothesis, but indicate that piano-based therapy requires greater than 2 weeks to begin improving dexterity and may influenced co-occurring socialization.

DETAILED DESCRIPTION:
The primary finding of this study is that older adults demonstrate improvements in manual dexterity after four weeks of piano training, but do not improve significantly after just two weeks. Furthermore, it does not matter whether the participants actively play for the first part and passively listen for the second part or vice versa.

Of the three proposed mechanisms of Music Supported Therapy (MST) explained in the introduction, the findings of this study may be best explained by the emotion-motivation mechanism. Though dexterity scores were organized by whether the scores followed an active playing module, all participants experienced the same amount of music-listening and social interaction. Whether the participant was playing the music him/herself or observing, both groups were always hearing the same songs and scales for the same amount of time. The emotion-motivation mechanism states that this music-listening alone may increase cognitive processes like working memory and boost both mood and motivation. Therefore, these findings may mean that listening to piano music helps dexterity performance in older adults; but it does so if and only if the participants experience the music-listening module for a sufficient duration of time.

Along with music-listening, social interaction was consistent between active and passive groups throughout the study. This interpersonal interaction may also have had an effect on mood and motivation, as piano instructors provided high levels of encouragement and complimented the participants' progress often. Relationship quality between patient and therapist is correlated with efficacy of therapy. This concept of increased socialization contributing to dexterity improvements is also supported by a study that identified social participation as a preventative factor of perceptual speed decline in older adults.

Not finding the hypothesized effect of active versus passive condition on dexterity could be due to dexterous activities that the participants were engaged in outside of the training modules. For example, three of the 15 participants reported that they currently play piano in their free time, so it can be conjectured that those participants were engaged in active piano playing even when they were in the passive listening module. Other activities enjoyed by participants include exercise classes and painting-both of which could have been improving or maintaining their dexterity throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Able to physically and cognitively withstand 30 minute piano training sessions

Exclusion Criteria:

-

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2017-10-21 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Purdue Pegboard | 10 minutes
  Fine Motor Manual Dexterity
Box and Block Test | 5 minutes
  Gross Motor Dexterity

CONTACTS AND LOCATIONS:
Locations (1):
- Shanango on the Green, New Wilmington, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
no identifiers. Confidential data.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately and for the next five years
Access Criteria: Researchers

REFERENCES:
- [Background] Ferreira PH, Ferreira ML, Maher CG, Refshauge KM, Latimer J, Adams RD. The therapeutic alliance between clinicians and patients predicts outcome in chronic low back pain. Phys Ther. 2013 Apr;93(4):470-8. doi: 10.2522/ptj.20120137. Epub 2012 Nov 8. PMID 23139428
- [Background] Jones L, Karageorghis CI, Ekkekakis P. Can high-intensity exercise be more pleasant?: attentional dissociation using music and video. J Sport Exerc Psychol. 2014 Oct;36(5):528-41. doi: 10.1123/jsep.2013-0251. PMID 25356615
- [Background] Lovden M, Ghisletta P, Lindenberger U. Social participation attenuates decline in perceptual speed in old and very old age. Psychol Aging. 2005 Sep;20(3):423-34. doi: 10.1037/0882-7974.20.3.423. PMID 16248702
- [Background] Vuilleumier P, Trost W. Music and emotions: from enchantment to entrainment. Ann N Y Acad Sci. 2015 Mar;1337:212-22. doi: 10.1111/nyas.12676. PMID 25773637